CLINICAL TRIAL: NCT00705718
Title: Endurant Stent Graft System US Clinical Study
Brief Title: Endurant Bifurcated and Aorto-Uni-Iliac (AUI) Stent Graft System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Medtronic - 089
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: Endurant Stent Graft System; Abdominal Aortic Aneurysms; Endovascular Treatment
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endurant Bifurcated arm (Experimental): The Bifurcated arm includes subjects who have received a bifurcated device. The Endurant Stent Graft System Bifurcated device is administered to treat patients with an Abdominal Aortic Aneurysm.
  Interventions: Device: Endurant Stent Graft System
- Endurant AUI arm (Experimental): The AUI arm includes subjects who have received an AUI device. The Endurant Stent Graft System AUI device is administered to treat patients with an Abdominal Aortic Aneurysm.
  Interventions: Device: Endurant Stent Graft System

INTERVENTIONS:
Device: Endurant Stent Graft System — Abdominal Aortic Aneurysm Repair
  Other Names: Endovascular treatment of Abdominal Aortic Aneurysm

SUMMARY:
To demonstrate safety and effectiveness of the Endurant Stent Graft in the treatment of Abdominal Aortic or Aorto-Uni-Iliac Aneurysms.

DETAILED DESCRIPTION:
Prospective, two-arm, non-randomized, multicenter clinical study enrolling subjects treated with the bifurcated stent graft in one arm and subjects treated with the AUI in a second arm.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old.
2. Subject (or Subject's legal representative) understands and voluntarily has signed and dated an Informed Consent document approved by the Sponsor and by the Institutional Review Board.
3. Subject is able and willing to comply with the protocol and undergo follow-up requirements.
4. Subject is a suitable candidate for elective surgical repair of AAA by as evaluated by American Society of Anesthesiologists (ASA) Physical Status Classification System I, II, III, or IV
5. Subject has an abdominal aortic or aortoiliac aneurysm characteristics that meet protocol parameter
6. Subject meets all the protocol anatomical criteria* as demonstrated on contrast-enhanced CT or MRA
7. Subject has vascular dimensions in the range of sizes available for the Endurant Stent Graft
8. Subject has documented imaging evidence of at least 1 patent iliac and 1 femoral artery, or can tolerate a vascular conduit that allows introduction of the device.
9. Subject's native vessel anatomy is more suited for the introduction and/ or deployment of an Endurant Uni-Iliac Stent Graft System.

Exclusion Criteria:

1. Subject has a life expectancy < 1 year
2. Subject is participating in another investigational drug or device study
3. Subject requires emergent aneurysm treatment
4. Subject is a female of childbearing potential in whom pregnancy cannot be excluded.
5. Subject has a known hypersensitivity or contraindication to anticoagulants, antiplatelets, or contrast media, which is not amenable to pre-treatment.
6. Subject is morbidly obese (body mass index ≥ 40 kg/m2) or has other documented clinical conditions that severely inhibit radiographic visualization of the aorta.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2016-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel S Makaroun, MD, Principal Investigator — Division of Vascular Surgery University of Pittsburgh Medical Center
Locations (30):
- United States (30):
  - University of Alabama Hospitals, Birmingham, Alabama
  - Arizona Heart Institute, Phoenix, Arizona
  - Stanford University Medical Center, Stanford, California
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Good Samaritan Hospital, Downers Grove, Illinois
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical Center, Albany, New York
  - Sisters of Charity Hospital, Buffalo, New York
  - NYU Hospitals Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Mission Hospitals, Asheville, North Carolina
  - Mid Carolina Presbyterian Hospital, Charlotte, North Carolina
  - Lindner Clinical Trial Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Jobst Vascular Center, Toledo, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sanford Research, Sioux Falls, South Dakota
  - Baptist Memorial Hospital Memphis, Memphis, Tennessee
  - Premier Surgical Associates, Powell, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Scott & White Memorial Medical Center, Temple, Texas
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Endurant AUI Arm: Endurant Stent Graft System : Abdominal Aorto-Uni-Iliac Aneurysm Repair
- Endurant Bifurcated Arm: Endurant Stent Graft System : Abdominal Aortic Aneurysm Repair
Period: Overall Study
Arm/Group | Endurant AUI Arm | Endurant Bifurcated Arm
Started | 44 | 150
1 Month Follow up | 43 (1 Death) | 149 (1 Subject Missed Visit)
6 Month Follow up | 40 (3 Deaths) | 143 (2 Deaths, 5 Subjects Missed Visit)
12 Month Follow up | 37 (2 Deaths) | 128 (4 Deaths, 12 Subjects Not due for next visit, 4 Subjects Missed Visit)
Completed | 37 | 128
Not Completed | 7 | 22
Not completed — Death | 6 | 6
Not completed — Not due for Visit | 0 | 12
Not completed — Follow up not done | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endurant AUI Arm | Endurant Bifurcated Arm | Total
Number analyzed (Participants) | 44 | 150 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (7.6) | 73.1 (8.0) | 73.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 30 | 137 | 167
Region of Enrollment [Number; unit: participants]
  United States | 41 | 150 | 191
  Canada | 3 | 0 | 3
Baseline Medical History [Number; unit: participants] — The Overall Number of Baseline Participants number may differ from the number within each baseline measure category. The Category number indicates the number of Participants with the baseline measure within that category.
  participants
    Angina | 11 | 27 | 38
    Arrhythmia | 15 | 59 | 74
    Congestive Heart Failure | 7 | 24 | 31
    Hypertension | 38 | 130 | 168
    Myocardial Infarction | 14 | 45 | 59
    Peripheral vascular disease | 33 | 34 | 67
    Abnormal renal function | 14 | 43 | 57
    Chronic obstructive pulmonary disorder | 26 | 53 | 79
    Diabetes | 11 | 40 | 51
    Tabacco use in the last 10 years | 29 | 66 | 95

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint (Freedom From MAEs Within 30 Days of Index Procedure)
Description: The primary safety endpoint is composite defined as the proportion of subjects free from major adverse events (MAE) within 1 month (day 0 - Day 30)of implant is non-inferior to the proportion of subjects free from MAEs in the Talent Control Group. The endpoint is defined as the proportion of subjects free from occurence of a MAE within 1 month of the implantation of the Endurant Stent Graft. The major adverse events composite endpoint which will be evaluated at 1 month post implant includes the occurrence of any of the following events.
  * All-Cause Mortality
  * Bowel Ischemia
  * Myocardial Infarction
  * Paraplegia
  * Procedural Blood Loss > or equal to 1000 cc
  * Renal Failure
  * Respiratory Failure
  * Stroke
Time Frame: 30 days (Safety)
Population: Freedom from Major Adverse Events within 30 Days of Implant
Measure: Number; unit: percentage of participants
Arm/Group | Endurant AUI Arm | Endurant Bifurcated Arm
Number analyzed (Participants) | 44 | 150
percentage of participants | 88.6 | 96.0

2. Primary Outcome: Major Adverse Events Within 30 Days of Index Procedure
Description: as for outcome 1
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | Endurant AUI Arm | Endurant Bifurcated Arm
Number analyzed (Participants) | 44 | 150
percentage of participants
  MAEs within 30 days | 11.4 | 4.0
  All Cause Mortality | 2.3 | 0
  Myocardial Infarction | 6.8 | 0.7
  Respiratory Failure | 4.5 | 1.3
  Paraplegia | 0 | 0
  Stroke | 2.3 | 0.7
  Bowel Ischemia | 0 | 1.3
  Procedural Blood Loss > or equal to 1000 cc | 4.5 | 0.7
  Renal Failure | 2.3 | 0.7

3. Secondary Outcome: Secondary Endpoints - Safety Evaluation
Description: The following secondary endpoints were included in the Pivotal trial to evaluate the safety profile of the Endurant Stent Graft System.
  * Aneurysm-Related Mortality through 12 months
  * All-Cause Mortality with 30 days
  * All-Cause Mortality within 12 months
  * Major Adverse Events through 12 months
  * Adverse Events through 12 months
  * Unanticipated Adverse Device Events
  * Serious Adverse Events (SAEs) As reported at the time of the data cut off.
  * Device Related Adverse Events
  * Procedure Related Adverse Events
  * Adverse Events (excluding SAEs)
Time Frame: 12 months
Population: Number of subjects enrolled in the study arm
Measure: Number; unit: percentage of evaluable participants
Arm/Group | Endurant AUI Arm | Endurant Bifurcated Arm
Number analyzed (Participants) | 44 | 150
percentage of evaluable participants
  Freedom from Aneurysm related Mortality through 12 | 100 | 100
  Freedom from All Cause Mortality through 30 Days | 97.7 | 100
  Freedom from All Cause Mortality through 12 months | 86.4 | 95.7
  Freedom from MAEs through 12 months | 72.7 | 89.2
  Serious Adverse Events through 12 months | 56.8 | 40.7
  Device Related Adverse Events through 12 months | 6.8 | 1.3
  Procedure Related AEs through 12 month | 70.5 | 58.0
  Adverse Events through 12 months | 90.9 | 80.0
  Unanticipated Adverse Events | 0 | 0.6

4. Primary Outcome: Primary Effectiveness Endpoint (Technical Success)
Description: Technical success defined as successful delivery and deployment of the stent graft in the planned location and with no unintentional coverage of both the internal iliac arteries or any visceral aortic branches and with removal of the system. Technical success was assessed intra-operatively.
Time Frame: Intra-operatively
Population: The Technical Success of the Endurant Bifurcated arm was based on obtaining information for the first 121 evaluable subjects available in the clinical study.
Measure: Number; unit: participants
Arm/Group | Endurant AUI Arm | Endurant Bifurcated Arm
Number analyzed (Participants) | 44 | 121
participants | 43 | 118

5. Primary Outcome: Primary Effectiveness Endpoint (Treatment Success)
Description: Treatment success is defined as Technical success and the following:
  * Freedom from AAA diameter increased, defined as >5 mm increase in maximum diameter as measured on CT scan (or MRA/MRI) at 12 months as compared to 1 month
  * Freedom from Types I and III endoleaks at 12 months including those requiring intervention through 12 months
  * Freedom from aneurysm rupture through 12 months
  * Freedom from conversion to surgery through 12 months
  * Freedom from stent graft migrations resulting in a serious adverse event or requiring secondary intervention through 12 months
  * Freedom from stent graft occlusion at 12 months
Time Frame: 12 months
Population: The number of evaluable subjects for ths endpoint.
Measure: Number; unit: participants
Arm/Group | Endurant AUI Arm | Endurant Bifurcated Arm
Number analyzed (Participants) | 36 | 121
participants
  Successful Aneurysm treatment | 35 | 118
  Type I or III Endoleaks through 12 months | 0 | 0
  Aneurysm Rupture through 12 months | 0 | 1
  Conversion to Surgery through 12 months | 0 | 0
  Stent Graft Migration through 12 months | 0 | 0
  Stent Graft occlusion at 12 months | 0 | 1

6. Secondary Outcome: Secondary Endpoint - Effectiveness Evaluation
Description: The following secondary endpoints were included in the pivotal trial to evaluate the effectiveness profile of the Endurant Stent Graft System.
  * Stent Graft migration through 12 months
  * Stent Graft Patency through 12 months
  * All stent Graft Endoleaks at 1-month, 6-months, and 12-month
  * Secondary Procedures to correct Type I and type III Endoleaks through 12 months
  * Secondary Endovascular Procedures through 12 months
  * Technical Observations through 12 months
Time Frame: 12 months
Population: Number of subjects enrolled in the study arm
Measure: Number; unit: percentage of evaluable subjects
Arm/Group | Endurant AUI Arm | Endurant Bifurcated Arm
Number analyzed (Participants) | 44 | 150
percentage of evaluable subjects
  Stent Graft Migration through 12m | 0.0 | 0.0
  Stent Graft Patency through 12m | 100.0 | 97.6
  All Stent Graft Endoleaks a 1m | 14.3 | 16.1
  All Stent Graft Endoleaks a 6m | 12.8 | 11.6
  All Stent Graft Endoleaks a 12m | 10.5 | 9.8
  Secondary Proced. for Type I & III endoleaks @ 12m | 0.0 | 0.0
  Secondary Procedures through 12m | 2.6 | 5.1
  Technical Observations through 12m | 10.8 | 3.9

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events are submitted by the clinical study sites via electronic Case Report Form and are then reviewed by the sponsor.
Groups:
- 1. Endurant AUI Arm: Endurant Stent Graft System - Endurant AUI arm
- 2. Endurant Bifurcated Arm: Endurant Stent Graft System - Endurant Bifurcated arm
Arm/Group | 1. Endurant AUI Arm | 2. Endurant Bifurcated Arm
Serious Adverse Events (participants affected / at risk) | 25/44 | 64/150
Other Adverse Events (participants affected / at risk) | 35/44 | 80/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Endurant AUI Arm (N=44) | 2. Endurant Bifurcated Arm (N=150)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Other Bleeding Complications (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 3 (3)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiopulmonary Failure (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 3 (3)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 2 (2)
New Arrhythmia (Cardiac disorders) | 1 (1) | 3 (3)
Other Cardiac Complications (Cardiac disorders) | 2 (2) | 2 (2)
Bowel Necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal Polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other Bleeding Complications (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other Bowel Complications (Gastrointestinal disorders) | 4 (4) | 4 (4)
Other Complications (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Chest Pain, Non-Cardiac (General disorders) | 0 (0) | 1 (1)
Death, Cause Unknown (General disorders) | 1 (1) | 0 (0)
Endoleak Type IIa (single patent collateral vessel) (General disorders) | 0 (0) | 1 (1)
Endoleak Type IIb (multiple patent collateral vessels) (General disorders) | 0 (0) | 1 (1)
Endoleak Type Ib (Distal end) (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 9 (9)
Multi-Organ Failure (General disorders) | 0 (0) | 1 (1)
Other Complications (General disorders) | 0 (0) | 8 (8)
Other Vascular Complications (General disorders) | 1 (1) | 1 (1)
Stenosis (General disorders) | 1 (1) | 1 (1)
Other Complications (Hepatobiliary disorders) | 1 (1) | 0 (0)
Other Bowel Complications (Infections and infestations) | 0 (0) | 1 (1)
Other Complications (Infections and infestations) | 0 (0) | 1 (1)
Other Renal Complications (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Septic Shock (Infections and infestations) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2)
Wound Infection (Infections and infestations) | 2 (2) | 1 (1)
Bleeding > 1000 cc, procedural (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Other Bleeding Complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Other Complications (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Other Renal Complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Other Vascular Complications (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Increased Creatinine (Investigations) | 0 (0) | 3 (3)
Other Bowel Complications (Investigations) | 0 (0) | 1 (1)
Other Complications (Investigations) | 1 (2) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Other Complications (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Other Pulmonary Complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other Orthopedic Complications (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other Vascular Complications (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Other Bowel Complications (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Other Renal Complications (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular Accident (CVA) - Stroke (Nervous system disorders) | 3 (3) | 3 (5)
Intra-Cranial/Cerebral Hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Other Complications (Nervous system disorders) | 0 (0) | 2 (2)
Other Neurological Complications (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Change In Mental Status (Psychiatric disorders) | 0 (0) | 2 (3)
Other Neurological Complications (Psychiatric disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Other Renal Complications (Renal and urinary disorders) | 1 (1) | 2 (2)
Other Urologic Complications (Renal and urinary disorders) | 1 (3) | 2 (2)
Renal Artery Stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 3 (3)
Other Vascular Complications (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Other Bleeding Complications (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other Complications (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other Pulmonary Complication (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Depression or Failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (4)
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aneurysm Rupture (Vascular disorders) | 0 (0) | 1 (1)
Embolism (non-pulmonary) (Vascular disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Other Cardiac Complications (Vascular disorders) | 0 (0) | 1 (1)
Other Vascular Complications (Vascular disorders) | 1 (1) | 3 (3)
Peripheral Ischemia (Vascular disorders) | 0 (0) | 1 (1)
Pseudoaneurysm (Vascular disorders) | 1 (1) | 0 (0)
Venous Insufficiency (Vascular disorders) | 0 (0) | 1 (1)
Vessel Rupture/Dissection (femoral, iliac, etc.) (Vascular disorders) | 2 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Endurant AUI Arm (N=44) | 2. Endurant Bifurcated Arm (N=150)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
New Arrhythmia (Cardiac disorders) | 0 (0) | 8 (10)
Other Cardiac Complications (Cardiac disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 16 (16)
Other Bowel Complications (Gastrointestinal disorders) | 0 (0) | 11 (12)
Fever (General disorders) | 7 (7) | 21 (21)
Other Complications (General disorders) | 0 (0) | 8 (8)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 8 (8)
Wound Infection (Infections and infestations) | 3 (3) | 0 (0)
Other Wound Complications (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 19 (20)
Low HCT/Low HGB (Investigations) | 3 (3) | 0 (0)
Other Complications (Investigations) | 0 (0) | 9 (9)
Other Complications (Metabolism and nutrition disorders) | 9 (11) | 9 (11)
Other Renal Complications (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (10)
Other Complications (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Other Complications (Nervous system disorders) | 6 (6) | 0 (0)
Other Neurological Complications (Nervous system disorders) | 6 (8) | 11 (12)
Other Complications (Psychiatric disorders) | 5 (5) | 0 (0)
Renal Insufficiency (Renal and urinary disorders) | 5 (5) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 3 (3) | 0 (0)
Other Pulmonary Complication (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0)
Other Complications (Skin and subcutaneous tissue disorders) | 8 (8) | 9 (9)
Hematoma (Vascular disorders) | 5 (5) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 9 (9)

LIMITATIONS AND CAVEATS:
Adverse Events and Serious Adverse Events listed in ClinicalTrials.gov were re-coded, using MeDRA codes. To do so, events were reclassified. As a result, data in listings may not match those in Clinical Update reports, SSEDs, or Instructions for Use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of single site experience is not allowed until the Multicenter results are published. The Multicenter manuscript will be made available to all authors & Medtronic prior to submission. Final analysis and review on the multicenter manuscript will require Medtronic approval.